CLINICAL TRIAL: NCT03686943
Title: Iatrogenic Drug Risk in People Over 75, With or Without Cognitive Disorders, From an Inventory of Their Family Pharmacy
Acronym: RIMPAP
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned project
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18 / RIMPAP; 2018-A02122-53 (Other: IdRCB)
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Elderly; Iatrogenic Drug Risk
Keywords: Elderly; Iatrogenic drug risk; Family pharmacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Patient over 75 years seen with the mobile extra hospital geriatric team
  Interventions: Other: Family pharmacy

INTERVENTIONS:
Other: Family pharmacy — Observation of the family pharmacy in elderly group

SUMMARY:
Many hospitalizations or emergency room visits are due to problems of iatrogenic medication, especially in elderly patients who are very often polymedicated. Moreover, they are more at risk because of fragility. This has an important socio-economic impact. It therefore seems important to act upstream of these adverse events and a review of the drugs available in the homes of elderly patients seems a good starting point.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 75 years with or without cognitive disorders

Exclusion Criteria:

* Refusal to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patient over 75 years seen with the mobile extra hospital geriatric team
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-28 (Estimated); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Iatrogenic drug risk in patients' homes | At the inclusion (baseline)
  Description of potential drug contraindications and potential unadvisable drug interactions highlighted from the analysis of the family pharmacy by Theriaque databased

CONTACTS AND LOCATIONS:
Overall Officials: Julie BOURGUEIL, MD, Principal Investigator — University Hospital, Tours